CLINICAL TRIAL: NCT03918473
Title: Effects of Mobilization Versus Manipulation on Function in Participants Reporting Chronic Ankle Instability
Brief Title: Effects of Mobilization Versus Manipulation on Function in Participants Reporting CAI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Cameron Bolton, Principal Investigator, Shenandoah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 668
Record Dates: First submitted 2019-04-02; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Ankle Sprains
Keywords: Functional Performance; Manual Therapy
MeSH Terms: conditions — Ankle Injuries | interventions — Movement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with Movement (Experimental): A weight- bearing mobilization directed to the talocrural joint in a standing position.
  Interventions: Other: Mobilization with Movement
- Thrust Mobilization (Experimental): A high velocity, low amplitude thrust mobilization directed to the talocrural joint with the participant in a non-weight bearing position.
  Interventions: Other: Thrust Mobilization

INTERVENTIONS:
Other: Mobilization with Movement — The MWM group will receive manual therapy with the following protocol: the participant will be relaxed and standing in a staggered stance with the involved foot on an eight-inch step and both feet facing forward. The clinician will be positioned in front of the participant's leg and a non-elastic belt will be placed around the distal leg of the participant and the clinician's pelvis. The clinician will then apply a sustained posteroanterior glide to the tibia through the belt by leaning backwards, while stabilizing the fixed talus and forefoot with both hands. The participant will perform a slow lunge until the end range of motion without their heel lifting off the ground. The belt will be kept perpendicular to the tibia throughout the movement and 2 sets of 10 repetitions will be applied.
  Arms: Mobilization with Movement
Other: Thrust Mobilization — The talocrural joint TM will be a high velocity low amplitude manual therapy technique. This technique will be applied with the participant in the supine position on a plinth. The clinician grasps the foot with one hand with the fifth finger contacting the anterior surface of the ankle at the talus. The other hand reinforces the contact points and both thumbs are placed on the sole of the participant's foot. The clinician gives slight caudal traction focused on the talocrural joint with the ankle dorsiflexed and everted. The therapist then applies a high-velocity thrust distraction technique to the talocrural joint. Only one thrust will be applied and no audible cavitation is required. This manual therapy technique will be performed once.
  Arms: Thrust Mobilization

SUMMARY:
The investigator's purpose is to compare the effects of talocrural joint mobilization with movement versus thrust mobilization on functional performance in subjects reporting chronic ankle instability (CAI).

DETAILED DESCRIPTION:
Joint mobilizations are reported to increase range of motion (ROM), postural control and proprioception, and decrease pain in individuals with CAI. However, there is no research comparing the effects of mobilization with movement (MWM) versus thrust mobilization (TM) directed at the talocrural joint on functional performance in this population.

Inclusion and exclusion criterion have been established utilizing the International Ankle Consortium guidelines. Using a convenience sampling, participants will be randomized into the MWM or TM group.

The MWM group will receive manual therapy with the following protocol: the participant will be relaxed and standing in a staggered stance with the involved foot on an eight inch step and both feet facing forward . The clinician will be positioned in front of the participant's leg and a non-elastic belt will be placed around the distal leg of the participant and the clinician's pelvis. The clinician will then apply a sustained posteroanterior glide to the tibia through the belt by leaning backwards, while stabilizing the fixed talus and forefoot with both hands. The participant will perform a slow lunge until the end range of motion without their heel lifting off the ground. The belt will be kept perpendicular to the tibia throughout the movement and 2 sets of 10 repetitions will be applied.

The talocrural joint TM will be a high velocity low amplitude manual therapy technique. This technique will be applied with the participant in the supine position on a plinth. The clinician grasps the foot with one hand with the fifth finger contacting the anterior surface of the ankle at the talus. The other hand reinforces the contact points and both thumbs are placed on the sole of the participant's foot. The clinician gives slight caudal traction focused on the talocrural joint with the ankle dorsiflexed and everted. The therapist then applies a high-velocity thrust distraction technique to the talocrural joint. Only one thrust will be applied and no audible cavitation is required. Each manual therapy technique will be performed once.

An examiner, who is blinded to involved limb and group allocation, will perform a baseline, immediate follow-up, and one-week follow-up examination of range of motion and functional performance. The participants will complete subjective outcome measures at baseline, immediately post intervention, and at 1 week post intervention including the Foot and Ankle Ability Measurement (FAAM), FAAM-Sport, and the Cumberland Ankle Instability Tool (CAIT). Participants will also complete baseline, immediate follow-up, and one-week follow up assessments of the Multiple Hop Test (MHT), three directions of the Star Excursion Balance test (SEBT), and weight bearing lunge test (WBLT).

Data analysis will be performed using International Business Machines Statistical Package for the Social Sciences (SPSS). Alpha level will be set p<0.05. Expecting to utilize separate 2 x 2 repeated measures analysis of variance (ANOVA) to assess changes in the FAAM, FAAM-Sport, CAIT, MHT, WBLT, and three directions of the SEBT.

ELIGIBILITY:
Criteria:

As adapted from the position statement from the International Ankle Consortium.

Inclusion Criteria:

* 18-35 years of age
* A history of at least 1 significant ankle sprain (The initial sprain must have occurred at least 12 months prior to study enrollment, associated with inflammatory symptoms (pain, swelling, etc), created at least 1 interrupted day of desired physical activity)
* The most recent injury must have occurred more than 3 months prior to study enrollment.
* A history of the previously injured ankle joint "giving way" and/or recurrent sprain and/or "feelings of instability."
* Cumberland Ankle Instability Tool (CAIT) < 24
* Foot and Ankle Ability Measure (FAAM)42: ADL scale < 90%, Sport scale < 80%

Exclusion Criteria:

* A history of previous surgeries to the musculoskeletal structures (i.e., bones, joint structures, nerves) in either limb of the lower extremity.
* A history of a fracture in either limb of the lower extremity requiring realignment
* Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months, which impacted joint integrity and function (i.e., sprains, fractures) resulting in at least 1 interrupted day of desired physical activity

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline Multiple Hop Test immediately after intervention and at 1 week follow-up. | Baseline, immediately after intervention, and 1 week
  The participants will hop between 10 pieces of white 2 x 2 cm tape. Participants will be instructed to hop once between each numbered marker and avoid any postural corrections. Participants will be allowed to progress if they were able to stand still keeping their hands on their hips at each marker. Three trials on each leg will be performed and amount of time to complete trial, number of fixed-support, and change-in-support balance strategies will be recorded. The average of the three trials will be taken.
Change in baseline weight bearing lunge test (WBLT) immediately after intervention and at 1 week follow-up. | Baseline, immediately after intervention, and 1 week
  Weight-bearing dorsiflexion range of motion (ROM) will be measured using the lunge test with a digital inclinometer (Acumar Single Digital Inclinometer Model ACU001) placed on a marked spot 15 cm below the base of the tibial tuberosity. Participants will place their hands on the wall and touch a vertical line with their knee, while keeping their knee in line with their second toe and their heel on the ground. Participants will perform three trials on either leg and the average of three test trials will be recorded.
Change in baseline Star Excursion Balance Test (SEBT) immediately after intervention and at 1 week follow-up. | Baseline, immediately after intervention, and 1 week
  Each participant is asked to maintain single-limb stance, with hands on their hips, while reaching in anterior, posteromedial, and posterolateral directions.
Change in baseline Foot and Ankle Ability Measure (FAAM)- Activities of Daily Living (ADL) Subscale immediately after intervention and at 1 week follow-up. | Baseline, immediately after intervention, and 1 week
  The FAAM- ADL is a 21-item tool that is designed to assess functional limitations related to foot and ankle conditions. Each item is scored on a Likert scale; 0 (unable to do) to 4 (no difficulty) and has total point value of 84 points, reported as a percent value.
Change in baseline Foot and Ankle Ability Measure (FAAM)- Sport subscale immediately after intervention and at 1 week follow-up. | Baseline, immediately after intervention, and 1 week
  The FAAM- Sport is a 7-item tool that is a sub-scale of the FAAM. Each item is scored on a Likert scale; 0 (unable to do) to 4 (no difficulty) with a total point value of 28 points, reported as a percent value.
Change in baseline Cumberland Ankle Instability Tool (CAIT) immediately after intervention and at 1 week follow-up. | Baseline, immediately after intervention, and 1 week
  9-item questionnaire that helps discriminate and measure the severity of functional ankle instability.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Bolton, PT, DPT, Principal Investigator — Shenandoah University Division of Physical Therapy
Locations (1):
- Shenandoah University, Winchester, Virginia, United States

REFERENCES:
- [Background] Gribble PA, Delahunt E, Bleakley CM, Caulfield B, Docherty CL, Fong DT, Fourchet F, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino W, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Athl Train. 2014 Jan-Feb;49(1):121-7. doi: 10.4085/1062-6050-49.1.14. Epub 2013 Dec 30. PMID 24377963